CLINICAL TRIAL: NCT06422481
Title: Non-invasive Measurement of Myocardial Work Using Transthoracic Echocardiography in Critically Ill Patients: the MYOLOAD Study
Brief Title: Echocardiographic Measurement of Myocardial Work
Acronym: MYOLOAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-PP-04
Record Dates: First submitted 2024-05-06; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Physiological Phenomena; Intensive Care Unit Syndrome
MeSH Terms: interventions — Hypodermoclysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluids (Experimental)
  Interventions: Other: Fluid administration
- Norepinephrine (Experimental)
  Interventions: Other: Norepinephrine administration or increase in norepinephrine dosage

INTERVENTIONS:
Other: Fluid administration — Patients will receive fluid administration (500 mL of saline over 30 minutes). The indication of fluid administration will be left to the discretion of the attending physician.
  Arms: Fluids
Other: Norepinephrine administration or increase in norepinephrine dosage — Patients will receive norepinephrine or norepinephrine dosage will be increased if necessary to achieve the appropriate mean arterial pressure level. The indication of norepinephrine administration or increase in norepinephrine dosage will be left to the discretion of the attending physician.
  Arms: Norepinephrine

SUMMARY:
Echocardiography is recommended for the hemodynamic management of patients with shock. Recently, a new echocardiographic method has been proposed that provides a non-invasive measurement of myocardial work incorporating different components, namely total myocardial work (GWI), constructive myocardial work (GCW), lost myocardial work (GWW) and effective myocardial work (GWE). Echocardiographic measurement of myocardial work takes into account both myocardial deformation and left ventricular afterload (estimated by measuring systolic blood pressure) and, unlike the measurement of left ventricular ejection fraction and global longitudinal strain, could be less dependent on cardiac load conditions, particularly left ventricular afterload. To date, non-invasive measurement of myocardial work has never been validated in critically ill patients, and no study has assessed the effects of different therapies (fluids administration, administration of norepinephrine) on the different components of myocardial work in patients admitted to intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Indication to fluid administration left to the discretion of the attending physician
* Indication to norepinephrine administration or increase in norepinephrine dosage left to the discretion of the attending physician.

Exclusion Criteria:

* Patients under protection.
* Patients with do not ressuscitate order.
* Patients with severe left-side or right-side valvulopathy.
* Patients with atrial fibrillation.
* Patients with ventricular aneuvrysm or severe regional wall motion abnormalities.
* Patients with a pacemaker.
* Patients' objections to the collection of their health data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility of echocardiographic measurement | through study completion, an average of 1 year
  The primary outcome will be assess by evaluating the proportion of patients in whom non-invasive echocardiographic measurement of myocardial work is obtained.

SECONDARY OUTCOMES:
measurement of myocardial by cardiac ultrasound during fluid administration | through study completion, an average of 1 year
  The measurement of myocardial work will be performed non-invasively by cardiac ultrasound.
  The secondary outcomes will be assess the impact of fluid administration on the different components of myocardial work. as follows:
  (i) fluid-induced changes in the different components of myocardial work, (ii) concordance between changes in myocardial work and changes in cardiac output induced by fluid administration (iii), the ability of the different components of myocardial work to predict fluid responsiveness.
measurement of myocardial by cardiac ultrasound norepinephrine administration | through study completion, an average of 1 year
  The measurement of myocardial work will be performed non-invasively by cardiac ultrasound.
  The secondary outcomes will be assess the impact of norepinephrine administration on the different components of myocardial work. as follows:
  (i) norepinephrine-induced changes in the different components of myocardial work, (ii) concordance between changes in myocardial work and changes in cardiac output induced by norepinephrine and (iii), the ability of the different components of myocardial work to predict fluid responsiveness.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de NICE ARCHET, Nice, CHU de Nice
  - CHU de NICE PASTEUR, Nice, CHU de Nice
  - Aphm Hopital La Timone, Marseille